CLINICAL TRIAL: NCT04291066
Title: Prospective Analysis of the Use of N-Acetylcysteine and Vitamins in the Treatment of TBI in Geriatric Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: HonorHealth Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1445221
Record Dates: First submitted 2019-12-06; First posted 2020-03-02 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Acetylcysteine; Minerals

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): oral N-acetyl cysteine and oral multivitamin tablets
  Interventions: Drug: N-Acetyl cysteine
- Non-Treatment (No Intervention): Routine Care

INTERVENTIONS:
Drug: N-Acetyl cysteine — Carbonyl scavenger and multi-vitamins with minerals to neutralize reactive carbonyl groups on the lipid aldehydes in patients with TBI
  Other Names: Multi-vitamins with minerals
  Arms: Treatment

SUMMARY:
This study will evaluate the administration of N-Acetyl-cysteine in combination with multi-vitamins/minerals in geriatric population (>60 years of age) who have experienced a traumatic brain injury.

DETAILED DESCRIPTION:
This study aims to determine the effect of supplemental N-acetyl cysteine and additional multi-vitamin/mineral therapy on somatic, cognitive, and emotional post-concussion symptoms as determined by the Rivermeade Post-concussion Questionnaire (RPQ) within 24 hours of admission, post injury day 7, and post injury day 30. The RPQ questionnaires will be given to patients older than 60 years, who have been evaluated by the HonorHealth John C. Lincoln Medical Center or Deer Valley Medical Center trauma service within 3 hours of sustaining a traumatic brain injury (TBI).

ELIGIBILITY:
Inclusion Criteria:

* 60 years or older
* present to emergency department within 3 hours of documented TBI

Exclusion Criteria:

* patients without TBI
* patients with a history of TBI greater than 3 hours prior to presentation
* patients under the age of 60
* currently enrolled in an ongoing research study
* patients who at baseline prior to the TBI, cannot participate in cognitive function testing (aphasia, severe dementia, non verbal; prior to TBI)
* Patients who are unable to tolerate PO medications within 3 hours of sustaining TBI.

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Determine improvement in somatic, cognitive, and emotional post-concussion symptoms as measured by the Rivermeade Post-concussion Questionnaire (RPQ) in treatment group vs non-treatment group. | 1 to 30 days post traumatic brain injury event
  Somatic, cognitive, and emotional post-concussion symptoms as measured by, RPQ scores within 24 hours of admission, post injury day 7, and post injury day 30. The scale goes based on a zero to 4 grading system. Zero equaling "not experienced at all" to 4 equaling "a severe problem".

SECONDARY OUTCOMES:
Severity of common post TBI symptoms | 1 to 30 days post traumatic brain injury event
  The severity of the five most common post TBI symptoms, including headache, nausea, sleep disturbance, poor concentration and forgetfulness/poor memory as measured by the scores of individual questions in the Rivermeade Post-concussion Questionnaire within 24 hours of admission, post injury day 7, and post injury day 30. Scale is 0 to 64

CONTACTS AND LOCATIONS:
Overall Officials: Ryab mcPherson, DO, Principal Investigator — HonorHealth Research Institute
Locations (2):
- United States (2):
  - HonorHealth John C. Lincoln Medical Center, Phoenix, Arizona
  - HonorHealth Deer Valley Medical Center, Phoenix, Arizona

IPD SHARING:
Plan to Share IPD: No
Results will be published in peer-reviewed journal

REFERENCES:
- [Derived] Mcpherson RA, Mangram AJ, Barletta JF, Dzandu JK. N -acetylcysteine is associated with reduction of postconcussive symptoms in elderly patients: A pilot study. J Trauma Acute Care Surg. 2022 Nov 1;93(5):644-649. doi: 10.1097/TA.0000000000003639. Epub 2022 Apr 8. PMID 35393384